CLINICAL TRIAL: NCT02380248
Title: Clinical Evaluation of Systane® Gel Drops on Corneal Staining in Indian Subjects With Dry Eye
Brief Title: Clinical Evaluation of Systane® Gel Drops in Dry Eye Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXI639-P001 (C-13-040)
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Polyethylene Glycols; Propylene Glycol; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systane (Experimental): Polyethylene Glycol, 0.4%, Propylene Glycol, 0.3% eye drops, 1 drop QID in each eye for 90 days
  Interventions: Other: Polyethylene Glycol, 0.4%, Propylene Glycol, 0.3% eye drops

INTERVENTIONS:
Other: Polyethylene Glycol, 0.4%, Propylene Glycol, 0.3% eye drops
  Other Names: Systane® Gel Drops

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Systane® Gel Drops in dry eye subjects following 90 days of QID (4 times/day) dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must give informed consent, and be willing and able to attend all study visits.
* Best-corrected visual acuity (BCVA) of ≥ 55 letters in each eye as measured by ETDRS (letters read method).
* Dry eye in both eyes diagnosed by an ophthalmologist.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, test positive on a pregnancy test, or breast-feeding.
* Any medical condition (systemic or ophthalmic) that may, in the opinion of the Investigator, preclude the safe administration of test article or safe participation in the study.
* Any contraindications or hypersensitivities to the study medications or their components.
* Ocular surgery (of any type, including PRK, LASIK, Epilasik, etc.) or ocular trauma requiring medical or pharmacological treatment within 1 year of Screening.
* Use of topical ocular prescription or non-prescription medications, RESTASIS or topical ocular steroids within 14 days of Screening.
* Chronic medications (over the counter, prescription, or vitamins) that have not been on a stable dose for at least 30 days prior to Screening.
* Contact lens wear within 1 week of Screening and/or unwillingness to discontinue contact lens wear for the duration of the study.
* Participation in any other clinical trial within 30 days prior to Screening.
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head, CTM, Med Affairs, Study Director — Alcon Laboratories Pvt Ltd (India); Sr. Clinical Manager, Global Trial Leadership, Study Director — Alcon, A Novartis Division
Locations (1):
- Contact Alcon India for Trial Locations, Karnataka, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 13 study centers in India.
Pre-assignment Details: Of the 207 enrolled, 6 subjects were exited as screen failures prior to treatment. In addition, 1 subject met the entry criteria, but discontinued prior to the first instillation of investigational product (IP). This reporting group includes all treated subjects (200).
Groups:
- Systane: Polyethylene Glycol, 0.4%, Propylene Glycol, 0.3% eye drops, 1 drop QID (4 times/day) in each eye for 90 days
Period: Overall Study
Arm/Group | Systane
Started | 200
Completed | 186
Not Completed | 14
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were exposed to investigational product (Safety Analysis Set).
Arm/Group | Systane
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 118
Corneal Staining [Mean (Standard Deviation); unit: units on a scale] — Corneal staining was assessed by the Investigator through slit-lamp examination and reported on a scale of 0-3, where 0=normal (no staining) and 3=severe (numerous coalescent macropunctate areas and/or patches), for the 5 quadrants of each eye. The scores at each visit were summed by eye for each subject. The overall corneal staining score for the subject at each visit was then computed as the average of the sum from both eyes. Thus, the overall scores ranged between 0-15 with higher scores reflecting more damage to the corneal surface. Population: This analysis population includes all enrolled subjects who had a baseline and at least 1 postbaseline assessment of corneal staining (Full Analysis Set). Number analyzed includes number of subjects with non-missing response.
  units on a scale
    number analyzed (Participants) | 190
    (all) | 5.7 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corneal Staining at All Study Time Points
Description: Corneal staining was assessed by the Investigator through slit-lamp examination and reported on a scale of 0-3, where 0=normal (no staining) and 3=severe (numerous coalescent macropunctate areas and/or patches), for the 5 quadrants of each eye. The scores at each visit were summed by eye for each subject. The overall corneal staining score for the subject at each visit was then computed as the average of the sum from both eyes. Thus, the overall scores ranged between 0-15 with higher scores reflecting more damage to the corneal surface.
Time Frame: Baseline (Day 0), Day 45, Day 90
Population: Full Analysis Set. Number analyzed includes number of subjects with non-missing response in specified category.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Systane
Number analyzed (Participants) | 190
units on a scale
  Change from baseline at Day 45 | -2.7 (0.14)
  Change from baseline at Day 90: number analyzed (Participants) | 185
  Change from baseline at Day 90 | -4.0 (0.16)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the time of informed consent for the duration of a subject's participation in the study (up to 90 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered an IP regardless of whether or not the event had a causal relationship with the IP. AEs were obtained through elicited and spontaneous comments from subjects and through observations by the Investigator.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- Systane: All subjects exposed to study treatment
Arm/Group | Pretreatment | Systane
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/200
Other Adverse Events (participants affected / at risk) | 0/207 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.